CLINICAL TRIAL: NCT03420664
Title: The Effects of Different Types of Ankle Immobilisation in the Micro- and Macrocirculation
Brief Title: Comparison of the Effects of Lower Limb Immobilisation With Cast and Orthosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Paul Ackermann, Primary Investigator, Karolinska University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SW2017-02-IMMOB
Record Dates: First submitted 2017-02-09; First posted 2018-02-05 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Venous Stasis; Deep Venous Thrombosis
Keywords: cast; orthosis; immobilisation; venous stasis; circulation
MeSH Terms: conditions — Varicose Ulcer; Venous Thrombosis

STUDY DESIGN:
Intervention Model Description: Research subjects receive lower limb immobilisation with cast and with orthosis alternatively, randomised so as subsequent persons begin with different modality.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cast immobilisation (Experimental): A below knee cast is applied in order to achieve ankle immobilisation for one hour
  Interventions: Device: Below knee cast
- Orthosis (VACOped) immobilisation (Experimental): A below knee orthosis which allows for ankle movement is applied for one hour.
  Interventions: Device: Orthosis VACOped

INTERVENTIONS:
Device: Orthosis VACOped — Orthosis for lower limb immobilisation
  Arms: Orthosis (VACOped) immobilisation
Device: Below knee cast — Below knee cast for lower limb immobilisation
  Other Names: Plastrer cast of Paris
  Arms: Cast immobilisation

SUMMARY:
In this study we are going to measure the blood flow in the lower limbs under cast immobilisation and also under mobilisation with an orthosis. The aim is to evaluate how the aforementioned modalities affect the blood flow and also to compare between the two.

DETAILED DESCRIPTION:
Background: Lower limb immobilisation, for example after an Achilles tendon rupture, is known to be a cause for DVT, partly due to blood stasis. VACOped is a weight-bearing orthosis with adjustable range of motion of the ankle which is used in our department in patients operated for Achilles tendon rupture.

Aim: To assess the effects of a) lower leg casting in equinus without loading and b) application of the aforementioned orthosis with full weight baring in blood flow and microcirculation in the lower limbs.

Study Plan: Ten healthy individuals are planned to be recruited for this study. Blood flow in the Right popliteal will be measured with vein before, 30 and 60 min after the application of the cast or orthosis (alternate order between consequent individuals) with Duplex Ultrasound. The orthosis will be set to allow for ankle plantarflexion restricted between 15 and 30 degrees. Tissue oxygen saturation in the lower limbs will also be measured using a somatic regional oxymetry modality, INVOS, with adhesive sensors applied on each leg above the soleus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals

Exclusion Criteria:

* Severe cardiovascular or renal disease causing pitting oedema
* Previous operation in the lower limbs affecting the vascular or lymphatic system
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-02-10 (Actual); Primary Completion 2024-12-24 (Estimated); Study Completion 2025-12-24 (Estimated)

PRIMARY OUTCOMES:
The difference of the effect on the lower limb circulation between cast and VACOped immobilisation | 2.5 hours
  Duplex ultrasound (blood flow) and INVOS (regional tissue mixed saturation)

SECONDARY OUTCOMES:
Lower limb macrocirculation under cast immobilisation | 1 hour
  Duplex ultrasound (blood flow)
Lower limb microcirculation under cast immobilisation | 1 hour
  INVOS (regional tissue mixed saturation)
Lower limb macrocirculation under orthosis mobilisation | 1 hour
  Duplex ultrasound (blood flow)
Lower limb microcirculation under orthosis mobilisation | 1 hour
  INVOS (regional tissue mixed saturation)

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska university Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Publishing an abstract on Reasearch Gate